CLINICAL TRIAL: NCT05353621
Title: Resilience and Acute Stress in Simulation : "SimStress"
Brief Title: Resilience and Acute Stress in Simulation
Acronym: SimStress
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 00010254 - 2022 - 052
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Stress, Professional; Resilience; Anaesthesiology; Simulation
MeSH Terms: conditions — Occupational Stress

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: VAS reported Stress — VAS reported Stress measurement during simulation

SUMMARY:
The objective is to study an association between the resilience developed by anesthesia professionals and the level of acute stress during a simulation session.

DETAILED DESCRIPTION:
This trial will take place at the Grenoble Alpes University Hospital. Volunteer anaesthetists, nurse anaesthetists, professionals or students will perform a simulation scenario. This scenario generates a high level of stress and focuses on medication errors, which is a good educational tool for the participants.

The simulation is performed in an available operating room with a dedicated anesthesia cart. In this environment, 17 error opportunities were created, i.e., factors that could contribute to the occurrence of a medication error. A person playing the role of the anesthesiologist will give instructions, leave the room, and return to interrupt the participant several times, which will contribute to the intensity of the stressor. The simulation will proceed as follows:

Briefing:

Welcome and explanation of the session. Collection of age, gender, number of years in anesthesia, number of previous simulation sessions, participation or not in stress management training. Presentation of the context and the anesthesiologist, then the participants evaluate their stress using the VAS (visual analog scale) Stress, which triggers the beginning of the scenario. Introduction of the setting and the anesthesiologist, then participants rate their stress using the VAS Stress scale, triggering the start of the scenario.

Scenario:

10 minutes in length. After the briefing, the anesthesiologist announces the imminent arrival of a patient with a suspected abdominal aortic aneurysm. The participant must quickly prepare a tray of medications. The scenario ends just prior to the patient's arrival, with the anesthesiologist presenting the stress VAS again for further evaluation.

Debriefing:

The participant completes a questionnaire about opportunities for detected errors, followed by a 15-minute debriefing after the simulation session.

For each participant, data regarding stress VAS, CD-RISC, PSS-10 and number of errors detected will be compared.

The primary objective is to analyze an association between resilience developed by anesthesia professionals and acute stress level.

The secondary objectives are to study the association between the resilience developed by the anesthesia professionals and the level of acute stress present immediately at the end of the simulation.

immediately at the end of the simulation. Measure the association between resilience (CDRISC 10) and performance (number of potential errors detected). Compare resilience and acute stress between different statuses (anesthesiologist, intern, nurse anesthetist, student nurse anesthetist).

ELIGIBILITY:
Inclusion Criteria:

* Accepts Healthy Volunteers

Exclusion Criteria:

* Participants who object to the use of their data for research purposes.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: physician anesthesiologist or anesthesia intern or nurse anesthetist or student nurse anesthetist
Sampling Method: Non-Probability Sample
Enrollment: 79 (Actual)
Dates: Start 2022-05-18 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Resilience | 15 Days after simulation
  Measurement of resilience by Connor-Davidson Resilience Scale 10 (CD RISC 10 from 0 to 40) in participants. A high score indicates better resilience.
Self-reported stress | just Before the scenario (at 0 minute )
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).

SECONDARY OUTCOMES:
Performance | just after the end of scenario (at 10 minute)
  Number of potential errors detected by participants on a post-simulation questionnaire with 23 questions. 18 potential errors are present on the 23 questions. Each correct answer counts as one point and each error removes one point. The maximum score is 18. (performance 0-18); a higher score indicates better performance.
resilience of anesthetists | 15 Days after simulation
  Average measure of physician anesthesiologists' resilience by the Connor-Davidson Resilience Scale 10 (CD RISC 10 from 0 to 40). Higher scores indicate greater resilience.
resilience of Resident in anaesthesia | 15 Days after simulation
  Average measure of Resident in anaesthesia resilience by the Connor-Davidson Resilience Scale 10 (CD RISC 10 from 0 to 40). Higher scores indicate greater resilience.
resilience of nurse anesthetist | 15 Days after simulation
  Average measure of nurse anesthetist resilience by the Connor-Davidson Resilience Scale 10 (CD RISC 10 from 0 to 40). Higher scores indicate greater resilience.
resilience of the student nurse anesthetist | 15 Days after simulation
  Average measure of the student nurse anesthetist resilience by the Connor-Davidson Resilience Scale 10 (CD RISC 10 from 0 to 40). Higher scores indicate greater resilience.
Self-reported stress | just after the end of scenario (at 10 minute )
  Stress level self reported by participants on visual analogical scale (VAS from 0 to 100); One end of the scale represents the maximum conceivable symptom strength (i. e., 100%), the other end no symptoms whatsoever (i. e., 0%).

CONTACTS AND LOCATIONS:
Overall Officials: Yoann Zafiriou, Principal Investigator — University Hospital, Grenoble; Julien Picard, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital Grenoble, Grenoble, France